CLINICAL TRIAL: NCT04741516
Title: A Phase IV, Dose Optimized, Open Label, Evaluation of the Effect Foquest® (Methylphenidate HCl Controlled Release) on Sleep in Children Aged 6-12 With Attention Deficit Hyperactivity Disorder
Brief Title: Evaluation of the Effect Foquest® on Sleep in Children Aged 6-12 With ADHD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: JPM van Stralen Medicine Professional (Other)
Collaborators: Purdue Pharma, Canada (Industry)
Responsible Party: Principal Investigator, Dr. Judy van Stralen, Principal Investigator, JPM van Stralen Medicine Professional
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RES 19-009
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Foquest; Attention Deficit Hyperactivity Disorder; Sleep; Sleep latency
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medication arm (Experimental)
  Interventions: Drug: Foquest

INTERVENTIONS:
Drug: Foquest — The drug being evaluated in this study is controlled release methylphenidate HCl control (Foquest®). Foquest® is a novel formulation of MPH developed by Purdue Pharma (Canada) and is approved in Canada for the treatment of ADHD in patients six years of age and older. Foquest® is the first methylphenidate product approved in Canada with an onset of action within one hour and a duration of action up to and including 16 hours (Wigal et al.2016). Foquest® is an ADHD treatment option for patients who require a rapid onset of action and extended duration of action

SUMMARY:
The purpose of this study is to evaluate the effect of Foquest® on sleep, using actigraphy and sleep diaries, in children aged 6-12 compared to baseline on no medication. Sleep difficulties, including prolonged sleep onset latency and decreased total sleep time have a significant negative impact on the functioning of children. In adults, sleep deprivation may result in drowsiness and yawning. However, in children, this may manifest as mood and behavioural disturbances which may even mimic the classic symptoms of ADHD; hyperactivity, poor impulse control, and inattention. This can in turn negatively affect the day to day activities of a child such as social interactions and learning. A meta-analysis in 2015 showed that stimulant medications impair sleep of children and adolescents. Some researchers have argued that stimulant medication may improve sleep. Importantly there appears to be heterogeneity in the effects of stimulant medication on sleep with some people sleeping better and some people worse after taking Foquest®. Although the randomized controlled trials done to date have demonstrated the efficacy and outlined the safety profile of Foquest, there remains some unanswered questions about the practical implications in the real-world setting. Some clinicians have raised the concern, for example, that the extended duration of Foquest, may have a negative impact on sleep. This study will evaluate the effect of Foquest® on sleep and particularly sleep latency and self and parent reported sleep restorative quality. This would be a novel study as there is no objective or subjective data on the effect of the Foquest® on sleep latency and total sleep time in children aged 6-12.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is a heterogeneous neurobehavioral disorder characterized by a persistent pattern of developmentally inappropriate inattentiveness, impulsivity, and hyperactivity. It is the most common pediatric neurobiological condition affecting approximately 5-7% of children worldwide.

Sleep difficulties, including prolonged sleep onset latency and decreased total sleep time have a significant negative impact on the functioning of children. This may manifest as mood and behavioural disturbances which may even mimic the classic symptoms of ADHD; hyperactivity, poor impulse control, and inattention. This can in turn negatively affect the day to day activities of a child such as social interactions and learning. A meta-analysis in 2015 showed that stimulant medications impair sleep of children and adolescents. Some researchers have argued that stimulant medication may improve sleep. Importantly there appears to be heterogeneity in the effects of stimulant medication on sleep with some people sleeping better and some people worse after taking Foquest®.

To date, seven pharmacokinetic studies of FOQUEST and six phase 3 clinical trials have been conducted. FOQUEST has demonstrated efficacy in the treatment of ADHD symptoms in double-blind, randomized clinical trials in children (aged 6 to 12), adolescents (aged 12 to 17) and adults (aged 18 or older). However, some clinicians have raised the concern that the extended duration of Foquest, may have a negative impact on sleep.

The purpose of this study is to evaluate the effect of Foquest® on sleep, using actigraphy and sleep diaries, in children aged 6-12 compared to baseline on no medication. This study will particularly evaluate the effect of Foquest® on sleep latency and self and parent reported sleep restorative quality. This would be a novel study as there is no objective or subjective data on the effect of the Foquest® on sleep latency and total sleep time in children aged 6-12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 6 to 12 years at the time of consent/assent.
2. Subject's parent or legally authorized representative (LAR) must be mentally and physically competent to provide informed consent and subject must be competent to provide assent and be able and willing to comply with the study protocol, including the number of visits and study duration.
3. Patient meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria for a diagnosis of ADHD combined presentation, inattentive presentation or hyperactive/impulsive presentation based on history.
4. Patient has a blood pressure measurement within 95th percentile for age, sex and height.
5. Patient and parent (LAR) are willing, able and likely to comply with the study procedures and restrictions within the protocol including wearing an actigraphic wrist device.

Exclusion Criteria:

1. Subject has sleep disorder breathing condition or another sleep disorder that may interfere with the interpretation of the study.
2. Subject has any condition that, in the opinion of the investigator, represent an inappropriate risk to the subject or may confound the interpretation of the study including subject being in an agitated state.
3. Subject has a true allergy to methylphenidate, history of serious adverse reactions to methylphenidate or be known to be non-responsive to methylphenidate. Non-response is defined as methylphenidate use at various doses for a phase of at least four weeks at each dose with little or no clinical benefit in the past 10 years.
4. Subject has a known history or presence of structural cardiac abnormalities, cardiovascular or cerebrovascular disease, serious heart rhythm abnormalities, syncope, tachycardia, cardiac conduction problems (such as clinically significant heart block or QT interval prolongation), exercise-related cardiac events including syncope and pre-syncope, clinically significant bradycardia or moderate to severe hypertension.
5. Subject has a history of seizure disorder (other than a single childhood febrile seizure occurring before the age of 3 years).
6. Subject has glaucoma, hyperthyroidism, thyrotoxicosis, advanced arteriosclerosis, or severe renal insufficiency.
7. Females of child-bearing potential (FOCP) who are pregnant, planning on becoming pregnant or breast feeding.
8. Subject is currently, or within the past 14 days, receiving MAO inhibitors.
9. Subject has a primary diagnosis of bipolar disorder, as assessed at visit.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in sleep onset latency | 8 weeks
  The Sleep Self Report - Child Form (SSR-C) was designed to measure five domains including sleep habits, problems falling asleep, sleep duration, night waking and daytime sleepiness.
  The wGT3X-BT is ActiGraph's flagship activity monitor, used by researchers around the world to capture and record continuous, high resolution physical activity and sleep/wake information.

SECONDARY OUTCOMES:
Executive Function | 8 weeks
  The Behaviour Rating Inventory of executive Function-Parent Form (BRIEF-P) is a 90 item parent completed questionnaire with a global executive composite score (GEC). GEC is reported as a t-score and a t-score of less than 65 is within normal limits.
ADHD Symptoms | 8 weeks
  Physician-rated scale ADHD Rating Scale IV (ADHD-RS-IV); 18-items; each item is rated in frequency level from 0 to 3, with a score of 0 meaning the item is displayed by the child "rarely or never" and a score of 4 is "very often"; total score ranges from 0 to 54. A higher score indicates more significant ADHD symptomatology.
Severity of Illness | 8 weeks
  The severity of illness using the Clinical Global Impression-Severity of Illness (CGI-S), a 7 point scale which is physician rated, with a score of 1 indicating "normal or not at all" and 7 indicating "extremely ill". A higher score indicates a higher severity illness.
Improvements of Subjects | 8 weeks
  The severity of illness using the Clinical Global Impression-Improvement of Illness (CGI-I), a 7 point scale which is physician rated To evaluate the change in functional impairment in subjects. A score of 1 indicates very much improved while a score of 7 indicates very much worse
Safety-Adverse events | 8 weeks
  Adverse events are recorded at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Judy van Stralen, MD, Principal Investigator — Center for Pediatric Excellence
Locations (1):
- Center for Pediatric Excellence, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Shakankiry HM. Sleep physiology and sleep disorders in childhood. Nat Sci Sleep. 2011 Sep 6;3:101-14. doi: 10.2147/NSS.S22839. Print 2011. PMID 23616721
- [Background] Kidwell KM, Van Dyk TR, Lundahl A, Nelson TD. Stimulant Medications and Sleep for Youth With ADHD: A Meta-analysis. Pediatrics. 2015 Dec;136(6):1144-53. doi: 10.1542/peds.2015-1708. PMID 26598454
- [Background] Faraone SV, Sergeant J, Gillberg C, Biederman J. The worldwide prevalence of ADHD: is it an American condition? World Psychiatry. 2003 Jun;2(2):104-13. PMID 16946911
- [Background] Chatoor I, Wells KC, Conners CK, Seidel WT, Shaw D. The effects of nocturnally administered stimulant medication on EEG sleep and behavior in hyperactive children. J Am Acad Child Psychiatry. 1983 Jul;22(4):337-42. doi: 10.1016/s0002-7138(09)60668-3. No abstract available. PMID 6875127
- [Background] Stein MA, Weiss M, Hlavaty L. ADHD treatments, sleep, and sleep problems: complex associations. Neurotherapeutics. 2012 Jul;9(3):509-17. doi: 10.1007/s13311-012-0130-0. PMID 22718078
- [Background] Wigal SB, Wigal T, Childress A, Donnelly GAE, Reiz JL. The Time Course of Effect of Multilayer-Release Methylphenidate Hydrochloride Capsules: A Randomized, Double-Blind Study of Adults With ADHD in a Simulated Adult Workplace Environment. J Atten Disord. 2020 Feb;24(3):373-383. doi: 10.1177/1087054716672335. Epub 2016 Oct 17. PMID 27756854